CLINICAL TRIAL: NCT01737710
Title: A Randomized Open Label Mechanistic Study in Atopic Dermatitis to Assess the Immunogenicity of Fluzone® Intradermal and Intramuscular Vaccines
Brief Title: Atopic Dermatitis Research Network (ADRN) Influenza Vaccine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Atopic Dermatitis Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAIT ADRN-05
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Dermatitis, Atopic
Keywords: Influenza Vaccines; Dermatitis; Injections, Intradermal; Injections, Intramuscular; Skin Diseases; Skin Diseases, Eczematous; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn; Skin Diseases, Genetic
MeSH Terms: conditions — Dermatitis, Atopic; Influenza, Human; Dermatitis; Skin Diseases; Skin Diseases, Eczematous; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Genetic Diseases, Inborn; Skin Diseases, Genetic | interventions — Influenza Vaccines; Injections, Intramuscular; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 92 Non-atopic controls vaccinated with Fluzone® Intradermal (Experimental): Non-atopic controls who will receive a single dose of the seasonal 2012-2013 Fluzone® Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
  Interventions: Biological: Fluzone® Intradermal Vaccine
- Moderate to severe AD vaccinated with Fluzone® Intradermal (Experimental): 92 moderate to severe atopic dermatitis participants who will receive a single dose of the seasonal 2012-2013 Fluzone® Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
  Interventions: Biological: Fluzone® Intradermal Vaccine
- Moderate to severe AD vaccinated with Fluzone® (Intramuscular) (Active Comparator): 92 moderate to severe atopic dermatitis participants who will receive a single dose of the seasonal 2012-2013 Fluzone® (Intramuscular) influenza vaccine from 0.5 mL single dose vials.
  Interventions: Biological: Fluzone® (Intramuscular) vaccine
- Non-atopic controls vaccinated with Fluzone® (Intramuscular) (Active Comparator): 20 non-atopic controls who will receive a single dose of the seasonal 2012-2013 Fluzone® (Intramuscular) influenza vaccine from 0.5 mL single dose vials.
  Interventions: Biological: Fluzone® (Intramuscular) vaccine
- Mild AD participants vaccinated with Fluzone® Intradermal (Experimental): 20 mild atopic dermatitis participants who will receive a single dose of the seasonal 2012-2013 Fluzone® Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
  Interventions: Biological: Fluzone® Intradermal Vaccine

INTERVENTIONS:
Biological: Fluzone® Intradermal Vaccine — A 0.1mL single-dose, in a latex-free, pre-filled microinjection system with an ultra-fine micro-needle. The active substance is prepared from influenza viruses propagated in embryonated chicken eggs. Fluzone® Intradermal is approved for use in persons 18 through 64 years of age and will be purchased from Sanofi Pasteur, Inc.
  Other Names: Influenza Virus Trivalent Vaccine (Types A and B) (Avian); Influenza Virus Vaccine, 2012-2013 Formula
  Arms: 92 Non-atopic controls vaccinated with Fluzone® Intradermal; Mild AD participants vaccinated with Fluzone® Intradermal; Moderate to severe AD vaccinated with Fluzone® Intradermal
Biological: Fluzone® (Intramuscular) vaccine — A 0.5 mL single-dose delivered via syringe using single-dose vials. The active substance is prepared from influenza viruses propagated in embryonated chicken eggs. Fluzone® for intramuscular injection is approved for persons 6 months and older and will be purchased from Sanofi Pasteur, Inc.
  Other Names: Influenza Virus Trivalent Vaccine (Types A and B) (Avian); Influenza Virus Vaccine, 2012-2013 Formula
  Arms: Moderate to severe AD vaccinated with Fluzone® (Intramuscular); Non-atopic controls vaccinated with Fluzone® (Intramuscular)

SUMMARY:
Atopic dermatitis, also called eczema, is a disease in which the skin is dry and scaly with severe itching. People who have atopic dermatitis often have complications from skin infections; these can include eczema herpeticum after herpes simplex virus infection or eczema vaccinatum after smallpox vaccination. People with atopic dermatitis may suffer from skin infections and may therefore respond differently to vaccinations.

A new flu vaccine which is injected into the skin instead of into muscle has recently been approved by the Food and Drug Administration for vaccination of the general population including patients with atopic dermatitis. This new vaccine has been shown to work as well as the vaccine which is injected into muscle when tested in people without atopic dermatitis. The main purpose of this study is to compare how people with atopic dermatitis respond to this new flu vaccine compared to non-atopic volunteers without atopic dermatitis. The second purpose is to look at how people with atopic dermatitis respond to the new vaccine which is injected into the skin compared to the vaccine which is injected into muscle.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the ADRN Registry study;
* Active, mild to severe AD (lesions present) with or without a history of eczema herpeticum or who are non-atopic as diagnosed using the ADRN Standard Diagnostic Criteria; and
* Willing to sign the informed consent form prior to initiation of any study procedure.

Exclusion Criteria:

* Pregnant or lactating. Women of child bearing potential must avoid becoming pregnant (use of an effective method of contraception or abstinence) for the duration of their participation in the study;
* Have a known allergy to any component of the Fluzone® Intradermal or Fluzone® (Intramuscular) vaccines, including egg protein, or have had a severe allergic reaction to a previous dose of any influenza vaccine;
* known or suspected congenital or acquired immunodeficiency or who have had immunosuppressive therapy (excluding steroids) such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months;
* Received systemic steroid therapy for 2 or more weeks at a dose ≥ 20 mg/day prednisone equivalent within 1 month prior to the day of vaccination or expect to receive within 3 weeks post-vaccination;
* Received a cumulative dose of inhaled and/or intranasally administered corticosteroids ≥ 880 mcg/day fluticasone equivalent for 2 or more weeks within 1 month prior to the day of vaccination or expect to receive within 3 weeks post-vaccination;
* A chronic illness, including but not limited to, cardiac, renal, or auto-immune disorders, or diabetes, at a stage that could interfere with study conduct or completion, based on the opinion of the Investigator. Asthma and underlying allergic conditions such as allergic rhinitis are not exclusionary;
* A neoplastic disease or any hematologic malignancy. Participants who have been disease free for at least six months will not be excluded;
* Participated in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the four weeks preceding the study vaccination or who plan to participate in another clinical trial during the present study period;
* Any skin disease other than AD that might compromise the stratum corneum barrier (e.g., bullous disease, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease);
* Received blood or blood-derived products that might interfere with the assessment of immune response in the past 3 months prior to vaccination or who plan to receive such products during the study period;
* Received previous vaccination (Fluzone® or another vaccine) against influenza in the past 6 months prior to vaccination;
* Received any other live vaccines within 4 weeks or inactivated vaccines within 2 weeks prior to study vaccination or who plan to receive any vaccination during the study period;
* Thrombocytopenia or bleeding disorder in the 3 weeks preceding vaccination;
* Personal or family history of Guillain-Barré Syndrome;
* A first degree relative already enrolled in the study;
* Determined to be ineligible based on the opinion of the Investigator.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 368 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, MD, PhD, Study Chair — National Jewish Health
Locations (5):
- United States (5):
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health & Science University, Protland, Oregon

REFERENCES:
- [Background] Leung DY, Gao PS, Grigoryev DN, Rafaels NM, Streib JE, Howell MD, Taylor PA, Boguniewicz M, Canniff J, Armstrong B, Zaccaro DJ, Schneider LC, Hata TR, Hanifin JM, Beck LA, Weinberg A, Barnes KC. Human atopic dermatitis complicated by eczema herpeticum is associated with abnormalities in IFN-gamma response. J Allergy Clin Immunol. 2011 Apr;127(4):965-73.e1-5. doi: 10.1016/j.jaci.2011.02.010. PMID 21458658
- [Background] Prymula R, Siegrist CA, Chlibek R, Zemlickova H, Vackova M, Smetana J, Lommel P, Kaliskova E, Borys D, Schuerman L. Effect of prophylactic paracetamol administration at time of vaccination on febrile reactions and antibody responses in children: two open-label, randomised controlled trials. Lancet. 2009 Oct 17;374(9698):1339-50. doi: 10.1016/S0140-6736(09)61208-3. PMID 19837254
- [Background] Pulendran B, Li S, Nakaya HI. Systems vaccinology. Immunity. 2010 Oct 29;33(4):516-29. doi: 10.1016/j.immuni.2010.10.006. PMID 21029962
- [Background] Schneider L, Weinberg A, Boguniewicz M, Taylor P, Oettgen H, Heughan L, Zaccaro D, Armstrong B, Holliday A, Leung DY. Immune response to varicella vaccine in children with atopic dermatitis compared with nonatopic controls. J Allergy Clin Immunol. 2010 Dec;126(6):1306-7.e2. doi: 10.1016/j.jaci.2010.08.010. PMID 20889193
- [Result] Leung DYM, Jepson B, Beck LA, Hanifin JM, Schneider LC, Paller AS, Monti K, David G, Canniff J, Lorenzo MG, Weinberg A. A clinical trial of intradermal and intramuscular seasonal influenza vaccination in patients with atopic dermatitis. J Allergy Clin Immunol. 2017 May;139(5):1575-1582.e8. doi: 10.1016/j.jaci.2016.12.952. Epub 2017 Feb 13. PMID 28209343
- [Derived] Jalbert E, Lussier S, Johnson MJ, Jepson B, Calatroni A, David G, Leung D, Weinberg A. Lower influenza-specific cell-mediated immune responses in individuals with atopic dermatitis compared with healthy controls. Hum Vaccin Immunother. 2020 Nov 1;16(11):2727-2735. doi: 10.1080/21645515.2020.1747374. Epub 2020 Apr 29. PMID 32347777
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Atopic Dermatitis Research Network (ADRN) website — https://www.nationaljewish.org/adrn/index

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 464 participants between the ages of 18 to 64 years were recruited and 368 of those participants were enrolled at 5 sites in the US between 10/2012 and 03/2013
Groups:
- Non-AD, Intradermal: Non-atopic dermatitis (AD) controls who received a single dose of the seasonal 2012-2013 Fluzone Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
- Moderate to Severe AD, Intradermal: Moderate to severe atopic dermatitis (AD) participants who received a single dose of the seasonal 2012-2013 Fluzone Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
- Moderate to Severe AD, Intramuscular: Moderate to severe atopic dermatitis (AD) participants who received a single dose of the seasonal 2012-2013 Fluzone (Intramuscular) influenza vaccine from 0.5 mL single dose vials.
- Non-AD, Intramuscular: Non-atopic dermatitis (AD) controls who received a single dose of the seasonal 2012-2013 Fluzone (Intramuscular) influenza vaccine from 0.5 mL single dose vials
- Mild AD, Intradermal: Mild atopic dermatitis (AD) participants who received a single dose of the seasonal 2012-2013 Fluzone Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
Period: Overall Study
Arm/Group | Non-AD, Intradermal | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular | Non-AD, Intramuscular | Mild AD, Intradermal
Started | 114 | 105 | 105 | 23 | 21
Completed | 112 | 101 | 102 | 23 | 21
Not Completed | 2 | 4 | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0
Not completed — Vaccinated in Error/Ineligible | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-AD, Intradermal | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular | Non-AD, Intramuscular | Mild AD, Intradermal | Total
Number analyzed (Participants) | 114 | 105 | 105 | 23 | 21 | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 4 | 0 | 1 | 7
  Between 18 and 65 years | 114 | 103 | 101 | 23 | 20 | 361
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.82 (11.96) | 35.11 (11.29) | 36.39 (12.04) | 34.30 (9.79) | 36.43 (14.14) | 36.65 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 58 | 60 | 12 | 10 | 207
  Male | 47 | 47 | 45 | 11 | 11 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 11 | 7 | 4 | 41
  Not Hispanic or Latino | 104 | 96 | 94 | 16 | 17 | 327
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 0 | 5
  Asian | 5 | 8 | 5 | 2 | 0 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 33 | 43 | 3 | 11 | 112
  White | 80 | 57 | 53 | 16 | 10 | 216
  More than one race | 3 | 5 | 2 | 0 | 0 | 10
  Unknown or Not Reported | 2 | 1 | 1 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 114 | 105 | 105 | 23 | 21 | 368
Seroprotected at Baseline - influenza B [Count of Participants; unit: Participants] — The number of participants that achieved seroprotection against influenza B at baseline prior to vaccination. Seroprotection is defined as having a serum hemagglutination-inhibition [HAI] antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza B. The goal of the study was to examine the immune response to influenza vaccination against influenza B. Participants who were already seroprotected against influenza B prior to vaccination were excluded from all relevant analyses for influenza B.
  Participants | 9 | 5 | 11 | 5 | 1 | 31
Seroprotected at Baseline - influenza H1N1 [Count of Participants; unit: Participants] — The number of participants that achieved seroprotection against influenza H1N1 at baseline prior to vaccination. Seroprotection is defined as having a serum hemagglutination-inhibition [HAI] antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H1N1. The goal of the study was to examine the immune response to influenza vaccination against influenza H1N1. Participants who were already seroprotected against influenza H1N1 prior to vaccination were excluded from all relevant analyses for influenza H1N1.
  Participants | 52 | 45 | 55 | 12 | 9 | 173
Seroprotected at Baseline - influenza H3N2 [Count of Participants; unit: Participants] — The number of participants that achieved seroprotection against influenza H3N2 at baseline prior to vaccination. Seroprotection is defined as having a serum hemagglutination-inhibition [HAI] antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H3N2. The goal of the study was to examine the immune response to influenza vaccination against influenza H3N2. Participants who were already seroprotected against influenza H3N2 prior to vaccination were excluded from all relevant analyses for influenza H3N2.
  Participants | 51 | 45 | 55 | 12 | 9 | 172

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza B
Description: The difference in the percent of participants that achieved seroprotection against influenza B at Day 28 between non-AD and moderate to severe AD participants, following a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine. Seroprotection is defined as having a serum hemagglutination-inhibition (HAI) antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza B. Participants who achieved seroprotection prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percent of participants who achieved seroprotection at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 post vaccination
Population: Subset of the per protocol population that were not seroprotected against influenza B at baseline. These participants received a full dose of vaccine, provided blood samples on Day 0 and Day 28, and had no major protocol deviations
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 96 | 102
percentage of participants | 34.4 | 22.5
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.082, Fisher Exact — Null hypothesis: no difference in the percent of participants that were seroprotected against influenza B at Day 28 between the two groups; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.92 to 3.55]

2. Primary Outcome: Seroprotection, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza H1N1
Description: The difference in the percentage of participants that achieved seroprotection against influenza H1N1 at Day 28 between non-AD and moderate to severe AD participants, following a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine. Seroprotection is defined as having a serum hemagglutination-inhibition (HAI) antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H1N1. Participants who achieved seroprotection prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroprotection at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: Subset of the per protocol population that were not seroprotected against influenza H1N1 at baseline. These participants received a full dose of vaccine, provided blood samples on Day 0 and Day 28, and had no major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 63 | 59
percentage of participants | 84.1 | 86.4
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.801, Fisher Exact — Null hypothesis: no difference in the percent of participants that were seroprotected against influenza H1N1 at Day 28 between the two groups; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.26 to 2.56]

3. Primary Outcome: Seroprotection, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza H3N2
Description: The difference in the percentage of participants that achieved seroprotection against influenza H3N2 at Day 28 between non-AD and moderate to severe AD participants, following a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine. Seroprotection is defined as having a serum hemagglutination-inhibition (HAI) antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H3N2. Participants who achieved seroprotection prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroprotection at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: Subset of the per protocol population that were not seroprotected against influenza H3N2 at baseline. These participants received a full dose of vaccine, provided blood samples on Day 0 and Day 28, and had no major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 59 | 60
percentage of participants | 84.7 | 73.3
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.177, Fisher Exact — Null hypothesis: no difference in the percentage of participants that were seroprotected against influenza H3N2 at Day 28 between the two groups; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.75 to 5.71]

4. Secondary Outcome: Fold-difference in Geometric Mean Serum Hemagglutination-inhibition (HAI) Antibody Titers, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza B
Description: The fold-difference (defined as a ratio to describe the change from baseline to Day 28) in geometric mean serum HAI antibody titers against influenza B between non-AD and moderate to severe AD participants, following a single dose of the seasonal 2012-2013 Fluzone Intradermal vaccine. A fold-difference of greater than 1 indicated an increase in HAI antibody titers against influenza B as a result of vaccination; therefore, higher numbers indicate a greater probability of avoiding disease if infected with influenza B. Participants who achieved seroprotection (which is defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza B) prior to vaccination were excluded from the analysis.
Time Frame: Day 28 post vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: HAI antibody titers
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 96 | 102
HAI antibody titers | 2.6 [2.0 to 3.2] | 2.0 [1.6 to 2.6]
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.092, ANCOVA — Null hypothesis: the fold differences in geometric mean titers against influenza B are not different between the two groups; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [0.96 to 1.61]

5. Secondary Outcome: Fold-difference in Geometric Mean Serum Hemagglutination-inhibition (HAI) Antibody Titers, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza H1N1
Description: The fold-difference (defined as a ratio to describe the change from baseline to Day 28) in geometric mean serum HAI antibody titers against influenza H1N1 between non-AD and moderate to severe AD participants, following a single dose of the seasonal 2012-2013 Fluzone Intradermal vaccine. A fold-difference of greater than or equal to 1 indicated an increase in HAI antibody titers against influenza H1N1 as a result of vaccination; therefore, higher numbers indicate a greater probability of avoiding disease if infected with influenza H1N1. Participants who achieved seroprotection prior to vaccination were excluded from the analysis, which is defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H1N1.
Time Frame: Day 28 post vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: HAI antibody titers
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 63 | 59
HAI antibody titers | 22.4 [12.8 to 39.3] | 37.7 [21.6 to 65.8]
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.103, ANCOVA — Null hypothesis: the fold differences in geometric mean titers against influenza H1N1 are not different between the two groups; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [0.32 to 1.11]

6. Secondary Outcome: Fold-difference in Geometric Mean Serum Hemagglutination-inhibition (HAI) Antibody Titers, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza H3N2
Description: The fold-difference (defined as a ratio to describe the change from baseline to Day 28) in geometric mean serum HAI antibody titers against influenza H3N2 between non-AD and moderate to severe AD participants, following a single dose of the seasonal 2012-2013 Fluzone Intradermal vaccine. A fold-difference of greater than or equal to 1 indicated an increase in HAI antibody titers against influenza H3N2 as a result of vaccination; therefore, higher numbers indicate a greater probability of avoiding disease if infected with influenza H3N2 Participants who achieved seroprotection prior to vaccination were excluded from the analysis, which is defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H3N2.
Time Frame: Day 28 post vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: HAI antibody titers
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 59 | 60
HAI antibody titers | 10.1 [6.2 to 16.4] | 9.7 [6.0 to 15.8]
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.895, ANCOVA — Null hypothesis: the fold differences in geometric mean titers against influenza H3N2 are not different between the two groups; Mean Difference (Final Values) = 1.04, 95% CI 2-sided [0.60 to 1.80]

7. Secondary Outcome: Seroprotection, Moderate to Severe Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intramuscular - Influenza B
Description: The difference in the percentage of moderate to severe AD participants that achieved seroprotection against influenza B at Day 28 between those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine and those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone (Intramuscular) vaccine. Seroprotection is defined as having a serum hemagglutination-inhibition (HAI) antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza B. Participants who achieved seroprotection prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroprotection at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 post vaccination
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Moderate to Severe AD, Intradermal: Moderate to severe atopic dermatitis (AD) participants received a single dose of the seasonal 2012-2013 Fluzone Intradermal influenza vaccine via a single-dose pre-filled microinjection system (0.1mL).
- Moderate to Severe AD, Intramuscular: Moderate to severe atopic dermatitis (AD) participants received a single dose of the seasonal 2012-2013 Fluzone (Intramuscular) influenza vaccine from 0.5 mL single dose vials.
Arm/Group | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular
Number analyzed (Participants) | 96 | 92
percentage of participants | 34.4 | 33.7
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Moderate to Severe AD, Intramuscular; Test type: Superiority or Other; p > 0.999, Fisher Exact — Null hypothesis: no difference in the percentage of participants that were seroprotected against influenza B at Day 28 between the two groups; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.54 to 1.97]

8. Secondary Outcome: Seroprotection, Moderate to Severe Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intramuscular - Influenza H1N1
Description: The difference in the percentage of moderate to severe AD participants that achieved seroprotection against influenza H1N1 at Day 28 between those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine and those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone (Intramuscular) vaccine. Seroprotection is defined as having a serum hemagglutination-inhibition (HAI) antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H1N1. Participants who achieved seroprotection prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroprotection at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular
Number analyzed (Participants) | 63 | 53
percentage of participants | 84.1 | 92.5
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Moderate to Severe AD, Intramuscular; Test type: Superiority or Other; p = 0.253, Fisher Exact — Null hypothesis: no difference in the percentage of participants that were seroprotected against influenza H1N1 at Day 28 between the two groups; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.09 to 1.63]

9. Secondary Outcome: Seroprotection, Moderate to Severe Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intramuscular - Influenza H3N2
Description: The difference in the percentage of moderate to severe AD participants that achieved seroprotection against influenza H3N2 at Day 28 between those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine and those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone (Intramuscular) vaccine. Seroprotection is defined as having a serum hemagglutination-inhibition (HAI) antibody titer of 1:40 or greater, which represents a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H3N2. Participants who achieved seroprotection prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroprotection at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular
Number analyzed (Participants) | 59 | 49
percentage of participants | 84.7 | 93.9
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Moderate to Severe AD, Intramuscular; Test type: Superiority or Other; p = 0.218, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.06 to 1.58]

10. Secondary Outcome: Seroconversion, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza B
Description: The difference in the percentage of participants that achieved seroconversion at Day 28 between non-AD and moderate to severe AD participants, following a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine. Seroconversion is defined as a 4-fold or greater increase in serum hemagglutination-inhibition [HAI] antibody titers against influenza B compared to baseline values, which represents the minimum intended effect of vaccination. Participants who achieved seroprotection, defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza B, prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroconversion at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 96 | 102
percentage of participants | 40.6 | 30.4
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.140, Fisher Exact — Null hypothesis: no difference in the percentage of participants that were seroconverted against influenza B at Day 28 between the two groups; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.84 to 2.94]

11. Secondary Outcome: Seroconversion, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe AD, Intradermal - Influenza H1N1
Description: The difference in the percentage of participants that achieved seroconversion at Day 28 between non-AD and moderate to severe AD participants, following a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine. Seroconversion is defined as a 4-fold or greater increase in serum hemagglutination-inhibition [HAI] antibody titers against influenza H1N1 compared to baseline values, which represents the minimum intended effect of vaccination. Participants who achieved seroprotection, defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H1N1, prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroconversion at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 63 | 59
percentage of participants | 85.7 | 88.1
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.791, Fisher Exact — Null hypothesis: no difference in the percentage of participants that were seroconverted against influenza H1N1 at Day 28 between the two groups; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.24 to 2.65]

12. Secondary Outcome: Seroconversion, Non-Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intradermal - Influenza H3N2
Description: The difference in the percentage of participants that achieved seroconversion at Day 28 between non-AD and moderate to severe AD participants, following a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine. Seroconversion is defined as a 4-fold or greater increase in serum hemagglutination-inhibition [HAI] antibody titers against influenza H3N2 compared to baseline values, which represents the minimum intended effect of vaccination. Participants who achieved seroprotection, defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H3N2, prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroconversion at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Non-AD, Intradermal
Number analyzed (Participants) | 59 | 60
percentage of participants | 76.3 | 73.3
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Non-AD, Intradermal; Test type: Superiority or Other; p = 0.833, Fisher Exact — Null hypothesis: no difference in the percentage of participants that were seroconverted against influenza H3N2 at Day 28 between the two groups; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.47 to 2.92]

13. Secondary Outcome: Seroconversion, Moderate to Severe Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intramuscular - Influenza B
Description: The difference in the percentage of moderate to severe AD participants that achieved seroconversion at Day 28 between those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine and those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone (Intramuscular) vaccine. Seroconversion is defined as a 4-fold or greater increase in serum hemagglutination-inhibition [HAI] antibody titers against influenza B compared to baseline values, which represents the minimum intended effect of vaccination. Participants who achieved seroprotection, defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza B, prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroconversion at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular
Number analyzed (Participants) | 96 | 92
percentage of participants | 40.6 | 47.8
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Moderate to Severe AD, Intramuscular; Test type: Superiority or Other; p = 0.378, Fisher Exact — [p-value comment as in outcome 10, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.40 to 1.38]

14. Secondary Outcome: Seroconversion, Moderate to Severe Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intramuscular - Influenza H1N1
Description: The difference in the percentage of moderate to severe AD participants that achieved seroconversion at Day 28 between those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine and those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone (Intramuscular) vaccine. Seroconversion is defined as a 4-fold or greater increase in serum hemagglutination-inhibition [HAI] antibody titers against influenza H1N1 compared to baseline values, which represents the minimum intended effect of vaccination. Participants who achieved seroprotection, defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H1N1, prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroconversion at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular
Number analyzed (Participants) | 63 | 53
percentage of participants | 85.7 | 88.7
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Moderate to Severe AD, Intramuscular; Test type: Superiority or Other; p = 0.783, Fisher Exact — [p-value comment as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.21 to 2.62]

15. Secondary Outcome: Seroconversion, Moderate to Severe Atopic Dermatitis (AD), Intradermal vs. Moderate to Severe Atopic Dermatitis, Intramuscular - Influenza H3N2
Description: The difference in the percentage of moderate to severe AD participants that achieved seroconversion at Day 28 between those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone Intradermal vaccine and those given a single dose (0.1mL) of the seasonal 2012 - 2013 Fluzone (Intramuscular) vaccine. Seroconversion is defined as a 4-fold or greater increase in serum hemagglutination-inhibition [HAI] antibody titers against influenza H3N2 compared to baseline values, which represents the minimum intended effect of vaccination. Participants who achieved seroprotection, defined as having a sufficient antibody amount to avoid disease in half of the individuals infected with influenza H3N2, prior to vaccination were excluded from the analysis. The goal was to examine whether there was a difference between the two groups in the percentage of participants who achieved seroconversion at Day 28 who were not seroprotected prior to vaccination.
Time Frame: Day 28 Post Vaccination
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular
Number analyzed (Participants) | 59 | 49
percentage of participants | 76.3 | 87.8
Statistical Analysis 1: Comparison: Moderate to Severe AD, Intradermal vs Moderate to Severe AD, Intramuscular; Test type: Superiority or Other; p = 0.143, Fisher Exact; Null hypothesis: no difference in the percentage of participants that were seroconverted against influenza H3N2 at Day 28 between the two groups; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.13 to 1.39]

ADVERSE EVENTS:
Time Frame: From start of the study through end of the study (up to Day 28 visit).
Description: Only adverse events that fit the following criteria have been collected:
  * Reactogenicity events of grade 3 or higher severity occurring between Day 0 and Day 7
  * Adverse events of grade 3 or higher severity through Day 28 visit
  * Serious adverse events through Day 28 visit
Arm/Group | Non-AD, Intradermal | Moderate to Severe AD, Intradermal | Moderate to Severe AD, Intramuscular | Non-AD, Intramuscular | Mild AD, Intradermal
Serious Adverse Events (participants affected / at risk) | 1/114 | 1/105 | 0/105 | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/114 | 0/105 | 1/105 | 0/23 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-AD, Intradermal (N=114) | Moderate to Severe AD, Intradermal (N=105) | Moderate to Severe AD, Intramuscular (N=105) | Non-AD, Intramuscular (N=23) | Mild AD, Intradermal (N=21)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-AD, Intradermal (N=114) | Moderate to Severe AD, Intradermal (N=105) | Moderate to Severe AD, Intramuscular (N=105) | Non-AD, Intramuscular (N=23) | Mild AD, Intradermal (N=21)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No